CLINICAL TRIAL: NCT01026064
Title: Utility of the Cantharidin-induced Skin Blister Assay for Evaluation of Anti-inflammatory Effects of Macrolides in Healthy Volunteers
Brief Title: Cantharidin-induced Skin Blister for Testing Anti-inflammatory Effects of Macrolides
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 112593
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Inflammation
Keywords: Macrolides; Inflammation; Azithromycin; Cantharidin induced skin blister model
MeSH Terms: conditions — Inflammation | interventions — Cantharidin; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Part C- Azithromycin (Experimental): 2 x 250 mg once daily over 3 days
  Interventions: Other: Cantharidin; Drug: Azithromycin
- Part C- Placebo (Placebo Comparator): Once daily over 3 days
  Interventions: Other: Cantharidin; Drug: Placebo

INTERVENTIONS:
Other: Cantharidin — Cantharone topical liquid containing 0.7% cantharidin (blistering agent) is applied as 25 µL of 0.1% cantharone solution in acetone
Drug: Azithromycin — Zithromax (250 mg oral capsule).
  Arms: Part C- Azithromycin
Drug: Placebo — Matching placebo
  Arms: Part C- Placebo

SUMMARY:
The purpose of this study is to investigate the utility of the cantharidin-induced skin blister assay for evaluation of the anti-inflammatory effects of macrolides in healthy male volunteers.

DETAILED DESCRIPTION:
The study will consist of 3 parts. Part A of the study will assess the feasibility of different cantharidin blister induction/sampling timepoints (challenge options) ranging from 16/16 hours to 48/48 hours, including the ability to evaluate the acute and resolving phase of acute inflammation. In Part A, 4 to 8 healthy male volunteers will be included. This will be followed by Part B (in up to 12 subjects), aimed to select the optimum challenge option based on the reproducibility of read-outs across two challenge sessions. This option will be applied in Part C in up to 24 subjects in order to evaluate the utility of the assay to demonstrate anti-inflammatory effects of a standard macrolide (azithromycin). Part C is designed as a double-blind, placebo-controlled, parallel group trial. Following the first cantharidin challenge and blister evaluation, subjects will be randomised in a 1:1 ratio to receive azithromycin or placebo. Skin blister induction and assessment will be repeated immediately after treatment completion and, potentially, approximately 3 weeks later. The inflammatory response to cantharidin and its modulation by azithromycin will be evaluated by total and differential cell counts in blister fluid, monocyte/macrophage phenotyping and the measurement of selected inflammation mediators in blister fluid and serum.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician.
* Male between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* The subject has a body weight of more than or equal to 50 kg and a BMI 18.5 to 30 kg/m2.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Subjects with very fair skin type.
* Presence on either forearm of tattoos, naevi, scars, keloids, hyperpigmentation, excessive hair or any skin abnormalities that may, in the opinion of the investigator, interfere with study assessments.
* Subjects with a history of keloids, skin allergy, hypersensitivity or contact dermatitis, including previous reactions to dressings to be used in the study.
* Subjects with a history of lymphangitis and/or lymphoedema.
* Subjects with a history of HIV infection, hepatitis B or C.
* A positive pre-study drug/alcohol screen.
* Use of prescription or non-prescription drugs, including ergot derivatives e.g. dihydroergotamine (Dihydergot), vitamins, herbal and dietary supplements (including St John's Wort) within whichever is the longer period of 14 days or 5 half-lives (if known) prior to the first challenge day, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within 56-day period.

For part C only:

* QTcB or QTcF >450 msec, based on average QTc value of triplicate ECGs obtained over a brief recording period, if the first measurement shows abnormal QTc value.
* History of sensitivity to azithromycin, macrolide/ketolide antibiotics or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-06-04 (Actual); Primary Completion 2009-11-27 (Actual); Study Completion 2009-11-27 (Actual)

PRIMARY OUTCOMES:
Tolerability and safety of cantharidin-induced skin blister assay (as determined by AEs, pain intensity, systemic inflammatory response, healing time, and cosmetic appearance of blister area) | Study duration
Total cell count, neutrophil count and monocyte/macrophage count in blister fluid. | Part C: end of treatment and potentially 3 weeks later

SECONDARY OUTCOMES:
Monocyte/macrophage phenotype in blister fluid. | Part C: end of treatment and potentially 3 weeks later
Inflammatory mediators in blister fluid. | Part C: end of treatment and potentially 3 weeks later
Markers of neutrophil activation. | Part C: end of treatment and potentially 3 weeks later
Inflammatory mediators in serum. | Part C: end of treatment and potentially 3 weeks later
PK parameters for azithromycin in plasma and whole blood following the last dose of azithromycin, as well as azithromycin concentration in PMNs and, if possible, in peripheral blood mononuclear cells at selected time points. | Part C: end of treatment and potentially 3 weeks later
Exploratory Outcome: Additional inflammatory mediators of interest may be determined. | Part C: end of treatment and potentially 3 weeks later

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Pene Dumitrescu T, Anic-Milic T, Oreskovic K, Padovan J, Brouwer KL, Zuo P, Schmith VD. Development of a population pharmacokinetic model to describe azithromycin whole-blood and plasma concentrations over time in healthy subjects. Antimicrob Agents Chemother. 2013 Jul;57(7):3194-201. doi: 10.1128/AAC.02430-12. Epub 2013 Apr 29. PMID 23629714
- See also: Results for study 112593 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/112593?search=study&search_terms=112593#rs